CLINICAL TRIAL: NCT00633230
Title: Effects of Sho-saiko-to, a Herbal Formula, in Reducing Viral Load in Hepatitis C
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding secured
Sponsor: University of Virginia (Other)
Responsible Party: Professor of Nursing and Director of the Center for the Study of Complementary and Alternative Therapies, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGT006; IRB-HSR #12957
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C Virus
Keywords: hepatitis C virus; complementary and alternative medicine; peginterferon alfa and ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — shosaiko-to

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): standardized herbal formula, Sho-saiko-to (SST): 3 capsules containing 700 mg of the SST herbal extract/capsule and 28 mg of the excipients, magnesium stearate and silicon dioxide/capsule 2 x day
  Interventions: Drug: standardized herbal formula, Sho-saiko-to (SST)
- 2 (Placebo Comparator): placebo capsules that look and smell identical to the active Sho-saiko-to (SST) capsules
  Interventions: Other: placebo capsule identical to the active herbal formula

INTERVENTIONS:
Drug: standardized herbal formula, Sho-saiko-to (SST) — 3 capsules containing 700 mg of the Sho-saiko-to (SST) herbal extract/capsule and 28 mg of the excipients, magnesium stearate, and silicon dioxide/capsule 2 x day
  Arms: 1
Other: placebo capsule identical to the active herbal formula — 3 placebo capsules 2 x day
  Arms: 2

SUMMARY:
The purpose of this study is to (1) determine the effects of the herbal formula Sho-saiko-to (SST) compared to placebo in treating hepatitis C virus (HCV) in persons who have not responded to the current conventional therapy (peginterferon alfa and ribavirin) or who have relapsed or in those for whom conventional therapy is contraindicated; (2) determine the influence that SST will have on participant reports of depression/sadness, fear and uncertainty related to the HCV disease progression, and renewal of hope in these individuals; and (3) collect preliminary data needed to examine feasibility, patient acceptance, and any potential limitations of the study.

DETAILED DESCRIPTION:
Persons infected with hepatitis C virus (HCV) suffer from multiple symptoms caused by both the disease and the current conventional treatment (peginterferon alfa and ribavirin) if they can tolerate the treatment or have no contraindications to taking it. Most HCV-infected individuals eventually develop chronic liver disease that may progress to complications such as hepatocellular carcinoma, hepatic decompensation, and cirrhosis. What is not known is whether or not modulation of the HCV disease using the standardized herbal formulation Sho-saiko-to (SST), 3 capsules containing 700 mg of the SST herbal extract/capsule and 28 mg of the excipients, magnesium stearate and silicon dioxide/capsule 2 times a day, over 12 weeks might reduce or prevent the prevalence and severity of liver deterioration and symptoms. Thus, the objectives of this project are to: (a) demonstrate quantitatively in a sample of persons infected with HCV expected SST treatment-driven changes in serum levels of liver enzymes, viral load, and CD4+ and CD8+ T-cell counts by longitudinal statistical modeling, and to correlate these to the severity of individual symptoms, liver enzyme levels, and CD4+ and CD8+ T-cells as measured at screening, 4, 8, and 12 weeks; (b) examine in vitro the response of a line of HCV-infected cells to the standardized herbal formulation; and (c) assess the mechanism by which the herbal formulation may affect the HCV-infected cells in vitro. Taken together, the clinical and laboratory components of the study should provide a strong test of our primary hypothesis that compared to placebo a standardized combined herbal formulation, SST, will reduce viral load, liver enzymes, and improve CD4+ and CD8+ T-cell counts in persons infected with HCV who did not respond or have relapsed after peginterferon alfa and ribavirin or in those for whom this conventional therapy is contraindicated. Our long-term objectives are to identify the basic mechanisms underlying chronic HCV infection-related cytokines and immune mediators and to provide a rationale for mechanism-driven SST disease treatment. Confirming the effect of SST in chronic HCV infection will create a foundation for a potentially supportive approach to managing HCV disease-related and treatment-related symptoms. Ability to reduce liver damage or even prevent the side effects of conventional therapy through the use of a standardized herbal formula, SST, would be of potential benefit to thousands of persons infected with HCV by providing an herbal treatment when the current conventional therapy is not effective or is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hepatitis C virus (HCV) genotype 1 with detectable HCV RNA >2000IU/mL at baseline assessment.
* Have relapsed after the standard care peginterferon alfa and ribavirin, or did not respond, or standard care peginterferon alfa and ribavirin contraindicated.
* Age 18 to 65 years
* Gender: male or female
* If female of childbearing potential (uterus has not been removed), willingness to use an approved form of birth control with male sexual partners through entire study and for 3 months after study completion
* Chest x-ray negative for pulmonary disease within 6 months of enrollment

Exclusion Criteria:

* Age < 18 or > 65 years.
* Currently on peginterferon alfa and ribavirin therapy, or have been on this therapy within the past 6 months.
* Currently taking monoamine oxidase inhibitors (MAOIs) for depression or have a serious mental illness.
* Diagnosed with cardiac disease, including severe heart failure, arrhythmia; significant kidney disease; asthma or other obstructive or restrictive pulmonary disease, interstitial pneumonitis and/or hypoxemia, leading to difficulty breathing or shortness of breath; immune-mediated disease (e.g., rheumatoid arthritis, vasculitis).
* Pulmonary function resulting in Forced Expiratory Volume (FEV1) at least 80% predicted.
* Confirmed diagnosis of TB.
* Infected with HIV, hepatitis A, B, D, E, or other viral blood infection (e.g., EBV, CMV)
* Taking anticoagulant therapy or have had anticoagulants within 30 days of enrollment
* Have taken antiviral medications within past 30 days
* Laboratory tests resulting in:
* platelet count ≤100,000/mm3
* serum bilirubin >1.5 g/dL
* Prothrombin Time-International Normalized Ratio (INR) >1.5
* albumin <3.4 g/dL
* hemoglobin <13 g/dL in men, <12 g/dL in women
* Absolute Neutrophil Count (ANC) <1.5 k/dL
* serum creatinine >1.5 mg/dL
* alanine transaminase (ALT) > 10 x baseline
* Hypertension (SBP > 140 or DBP >90)
* Hypokalemia (K < 3.5)
* Liver biopsy results that reveal stage 4 fibrosis (cirrhosis)
* Cirrhosis or at risk for developing hepatocellular carcinoma as evidenced by an elevated AFP test at screening.
* Undergone transplant of any kind and/or taking corticosteroids or other immunosuppressive therapy (or have taken immunosuppressive therapy within the previous 6 months)
* Consuming alcohol.
* Hypersensitivity to any of the 7 components of SST.
* Taking over-the counter products that could potentially interact with the components of SST.
* Have participated in another investigational drug study within the past 60 days.
* Taking anthraquinone drugs or herbs containing anthraquinone
* In a methadone maintenance program.
* Using recreational drugs.
* Pregnant, breastfeeding, or unwillingness to use an approved form of birth control for women of childbearing potential.
* Unable to understand the consent process or study-related questions due to language barriers, cognitive impairment, or other reasons.
* Weigh more than 275 pounds, which could complicate liver biopsy procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Reduction in HCV viral load, improvement in liver enzymes (ALT and AST), improvement in CD4+ and CD8+ T-cell counts. | At 4, 8, 12, 16 weeks.

SECONDARY OUTCOMES:
Improvement in symptoms of depression/sadness, fear related to HCV disease progression, uncertainty, and hopelessness over time | At baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ann G Taylor, EdD, Principal Investigator — University of Virginia; Abdullah M Al-Osaimi, MD, Study Director — University of Virginia